CLINICAL TRIAL: NCT03581786
Title: A Phase III, Randomized, Placebo Controlled, Multicenter, Double-Blind Study Comparing Toripalimab Injection (JS001) Combined With Chemotherapy Versus Placebo Combined With Chemotherapy for Recurrent or Metastatic Nasopharyngeal Cancer
Brief Title: The Efficacy and Safety Study of TORIPALIMAB INJECTION Combined With Chemotherapy for Nasophapyngeal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-015-III-NPC
Record Dates: First submitted 2018-06-05; First posted 2018-07-10 (Actual); Results first posted 2022-04-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-08

CONDITIONS: Recurrent or Metastatic NPC
MeSH Terms: conditions — Recurrence | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo combine with chemotherapy (Placebo Comparator): Gemcitabine 1000 mg/m² IV are given on Days 1 & 8, and cisplatin 80 mg/m² IV are given on Day 1 of each cycle，placebo will be administered at the dose of 240 mg Q3W before that. Chemotherapy is given Q3W for up to 6 cycles and placebo for up to 2 years
  Interventions: Drug: Placebos
- TORIPALIMAB INJECTION(JS001 )combine with chemotherapy (Experimental): Gemcitabine 1000 mg/m² IV are given on Days 1 & 8, and cisplatin 80 mg/m² IV are given on Day 1 of each cycle，JS001 will be administered at the dose of 240 mg Q3W before that. Chemotherapy is given Q3W for up to 6 cycles and JS001 for up to2years
  Interventions: Biological: TORIPALIMAB INJECTION(JS001 ) combine with chemotherapy

INTERVENTIONS:
Biological: TORIPALIMAB INJECTION(JS001 ) combine with chemotherapy — TORIPALIMAB INJECTION(JS001 ) combine with chemotherapy
  Arms: TORIPALIMAB INJECTION(JS001 )combine with chemotherapy
Drug: Placebos — placebo combine with chemotherapy
  Arms: placebo combine with chemotherapy

SUMMARY:
This is a randomized, placebo-controlled, multi-center, double blinded, Phase III study to determine the efficacy and safety of TORIPALIMAB INJECTIO（JS001） in combination with gemcitabine/cisplatin compared with placebo in combination with gemcitabine/cisplatin as first-line treatment in patients with histological/cytological confirmation of recurrent or metastatic NPC. The primary endpoint is PFS in all patients. Approximately 280 patients who fulfill all of the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to one of the two treatment arms. patients will be randomly assigned to the combination of JS001 (Arm A) or placebo (Arm B) with gemcitabine and cisplatin given every 3 weeks (Q3W) in 3-week cycles.

DETAILED DESCRIPTION:
Total 289 patients were enrolled and randomized in a 1:1 ratio to the group of JS001 (Arm A) with gemcitabine and cisplatin or placebo (Arm B) with gemcitabine and cisplatin every 3 weeks (Q3W) in the 'during chemotherapy' phase. During the 'post-chemotherapy' phase, patients randomized to Arm A or Arm B will continue treatment with JS001 or placebo as maintenance therapy Q3W until excessive toxicity or progressive disease, withdrawal of consent or Investigator's judgement or a maximum of 2 years. Tumor evaluation scans will be performed at screening (as baseline) then every 6weeks in the first 12 months then every 9 weeks thereafter until objective disease progression. The primary objective is to compare PFS as assessed by the IRC in ITT population (all randomized patients).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years and ≤75 years.
* 2. Histological/cytological confirmation of NPC.
* 3. Primarily metastatic (stage IVB as defined by the International Union against Cancer and American Joint Committee on Cancer staging system for NPC, eighth edition) or recurrent NPC that is not amenable for local regional treatment or curative treatment.
* 4. At least 1 measurable lesion according to RECIST version 1.1.
* 5. Life expectancy ≥ 3 months

Exclusion Criteria:

* 1. History of severe hypersensitivity reactions to other mAbs or any ingredient of JS001.
* 2. Prior therapy targeting PD-1 receptor, or its ligand PD-L1, or cytotoxic T lymphocyte associated protein 4 (CTLA4) receptor.
* 3. Major surgical procedure other than for diagnosis of NPC within 28 days prior to randomization or anticipation of need for a major surgical procedure during the study
* 4. History of hypersensitivity to gemcitabine or cisplatin or to any of the excipients.
* 5. Female patients who are at pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (32):
- China (25):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangzhou
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangzhou
  - The Fifth Affiliated Hospital Sun Yat-Sen University - Medical Oncology, Zhuhai, Guangzhou
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital (Hainan Province People's Hospital), Haikou, Hainan
  - Hebei Oncology Hospital, Shijiazhuang, Hebei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & TechnologyTongji Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Oncology Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Singapore (2):
  - National Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - TaiChung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi Y, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Wang S, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Luo X, Wang X, Tang X, Feng H, Yao S, Keegan P, Xu RH. Toripalimab Plus Chemotherapy for Recurrent or Metastatic Nasopharyngeal Carcinoma: The JUPITER-02 Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1961-1970. doi: 10.1001/jama.2023.20181. PMID 38015220
- [Derived] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Combine With Chemotherapy: In the during-chemotherapy phase, placebo will be given before gemcitabine and cisplatin, placebo will be administered at the dose of 240 mg Q3W,gemcitabine 1000 mg/m² IV over 30 minutes are given on Days 1 & 8, and cisplatin 80 mg/m² IV over 4 hours are given on Day 1 of each cycle. Chemotherapy is given Q3W for up to 6 cycles.
  During the post-chemotherapy phase, placebo and best supportive care (BSC) can be continued Q3W until excessive toxicity or progressive disease, withdrawal of consent, at the discretion of the Investigator or for a maximum of 2 years.
- TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy: In the during-chemotherapy phase, JS001 will be given before gemcitabine and cisplatin, JS001 will be administered at the dose of 240 mg Q3W,gemcitabine 1000 mg/m² IV over 30 minutes are given on Days 1 & 8, and cisplatin 80 mg/m² IV over 4 hours are given on Day 1 of each cycle. Chemotherapy is given Q3W for up to 6 cycles .
  During the post-chemotherapy phase, JS001 and best supportive care (BSC) can be continued Q3W until excessive toxicity or progressive disease, withdrawal of consent, at the discretion of the Investigator or for a maximum of 2 years.
Period: Overall Study
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Started | 143 | 146
Completed | 67 | 89
Not Completed | 76 | 57
Not completed — Death | 67 | 47
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 7 | 4
Not completed — reason other than specified above | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy | Total
Number analyzed (Participants) | 143 | 146 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 136 | 139 | 275
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.68 (10.355) | 45.84 (11.26) | 47.74 (10.973)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 116 | 124 | 240
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 143 | 146 | 289
Region of Enrollment [Number; unit: participants]
  Singapore | 2 | 3 | 5
  China | 134 | 136 | 270
  Taiwan | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: IRC-assessed Progression-Free Survival (PFS) According to RECIST v1.1
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy as measured by IRC-assessed progression free survival (PFS) according to RECIST v1.1 in all patients.
  The definition of Progressive Disease: At least a 20% increasein the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. or the appearance of one or more new lesions is also considered progression.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
months | 8.2 [7.03 to 9.79] | 21.4 [11.73 to NA] — Due to insufficient number of participants with events, the upper limit of the survival curve hasn't reached 50%, there is no estimate for the upper confidence limit on the median.

2. Secondary Outcome: OS
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: The time frame of OS collected is upto about 48months.
Population: NE below means "not estimable".
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
months | 33.7 [27.01 to 44.19] | NA [38.70 to NA] — Due to insufficient number of participants with events, median and the upper limit of the survival curve hasn't reached 50%, there is no estimate for the median and the upper confidence limit on the median.

3. Secondary Outcome: Investigator-assessed ORR According to RECIST v1.1
Description: To evaluate the efficacy of TORIPALIMAB INJECTION(JS001) plus chemotherapy compared with placebo plus chemotherapy, as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1.
Time Frame: From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 75.5 [67.64 to 82.32] | 82.2 [75.01 to 88.02]

4. Secondary Outcome: Investigator-assessed DoR According to RECIST v1.1
Description: To evaluate the efficacy of TORIPALIMAB INJECTION(JS001 )plus chemotherapy compared with placebo plus chemotherapy, as measured by investigator-assessed duration of response (DoR) according to RECIST v1.1.
Time Frame: From date of response until progressive disease. Up to 2 approximately years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 108 | 120
months | 6.0 [5.75 to 7.16] | 16.0 [11.93 to 22.47]

5. Secondary Outcome: Investigator-assessed DCR According to RECIST v1.1
Description: To evaluate the efficacy of TORIPALIMAB INJECTION(JS001) plus chemotherapy compared with placebo plus chemotherapy, as measured by investigator-assessed disease control rate (DCR) according to RECIST v1.1.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 90.9 [84.96 to 95.07] | 91.1 [85.26 to 95.17]

6. Secondary Outcome: Investigator-assessed PFS According to RECIST v1.1
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by Investigators-assessed PFS according to RECIST v1.1
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
months | 8.1 [7.10 to 8.61] | 17.3 [13.34 to 23.26]

7. Secondary Outcome: Investigator-assessed PFS Rate at 1 Year
Description: To evaluate the PFS rate at 1 year in each treatment arm by investigator
Time Frame: up to approximately 1years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 26.2 [18.96 to 33.99] | 61.4 [52.28 to 69.27]

8. Secondary Outcome: OS Rate at 1 Year
Description: To evaluate the OS rate at 1 year in each treatment arm
Time Frame: Up to approximately 1 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 87.1 [80.36 to 91.69] | 90.9 [84.87 to 94.62]

9. Secondary Outcome: IRC-assessed ORR According to RECIST v1.1
Description: health related quality of life (HRQoL) in patients treated with JS001 plus chemotherapy compared with placebo plus chemotherapy using the EORTC QLQ-H&N35
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 67.1 [58.79 to 74.75] | 78.8 [71.24 to 85.09]

10. Secondary Outcome: IRC-assessed DoR According to RECIST v1.1
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by IRC-assessed duration of response (DoR) according to RECIST v1.1.
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 96 | 115
months | 6.0 [5.55 to 8.25] | 18.0 [10.51 to NA] — Due to insufficient number of participants with events, the upper limit of the survival curve has not reached 50%, there is no estimate for the upper confidence limit on the median.

11. Secondary Outcome: IRC-assessed DCR According to RECIST v1.1
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by IRC-assessed disease control rate (DCR) according to RECIST v1.1.
Time Frame: From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 80.4 [72.96 to 86.58] | 88.4 [82.01 to 93.07]

12. Secondary Outcome: Number of Participants Experiencing an Adverse Event(AE)
Description: Incidence of adverse events(AE) as assessed by CTCAE version 5.0
Time Frame: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Participants | 143 | 146

13. Secondary Outcome: Anti-drug Antibody(ADA)
Description: To evaluate the incidence of ADAs against JS001
Time Frame: as for outcome 3
Population: ADA testing only was applicable for Toripalimab group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 0 | 146
Participants | 0 | 10

14. Secondary Outcome: PFS IRC-assessed Per irRECIST
Description: To evaluate PFS of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
months | 8.3 [7.06 to 9.89] | 21.6 [13.17 to NA] — Due to insufficient number of participants with events, the upper limit of the survival curve has not reached 50%, there is no estimate for the upper confidence limit on the median.

15. Secondary Outcome: ORR IRC-assessed Per irRECIST
Description: To evaluate ORR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 67.8 [59.51 to 75.39] | 78.8 [71.24 to 85.09]

16. Secondary Outcome: DoR IRC-assessed Per irRECIST
Description: To evaluate DoR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: From date of response until progressive disease. Up to 2 approximately years
Population: NE below means "not estimable"
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 97 | 115
months | 5.9 [5.55 to 8.25] | 20.1 [14.09 to NA] — Due to insufficient number of participants with events, the upper limit of the survival curve has not reached 50%, there is no estimate for the upper confidence limit on the median.

17. Secondary Outcome: DCR IRC-assessed Per irRECIST
Description: To evaluate DCR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 81.8 [74.51 to 87.77] | 88.4 [82.01 to 93.07]

18. Secondary Outcome: Investigator-assessed PFS Rate at 2 Years
Description: To evaluate the PFS rate at 2 years in each treatment arm by investigator
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 15.4 [9.59 to 22.53] | 37.0 [26.53 to 47.43]

19. Secondary Outcome: OS Rate at 2 Years
Description: To evaluate the OS rate at 2 years in each treatment arm
Time Frame: Up to approximately 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 65.1 [56.50 to 72.44] | 78.0 [70.18 to 83.97]

20. Secondary Outcome: PFS Investigator-assessed Per irRECIST
Description: To evaluate PFS of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
months | 8.1 [7.06 to 8.61] | 17.3 [13.34 to 23.26]

21. Secondary Outcome: ORR Investigator-assessed Per irRECIST
Description: To evaluate ORR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 75.5 [67.64 to 82.32] | 82.2 [75.01 to 88.02]

22. Secondary Outcome: DoR Investigator-assessed Per irRECIST
Description: To evaluate DoR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: From date of response until progressive disease. Up to 2 approximately years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 108 | 120
months | 5.9 [5.72 to 7.16] | 16.0 [11.93 to 22.47]

23. Secondary Outcome: DCR Investigator-assessed Per irRECIST
Description: To evaluate DCR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST.
Time Frame: Up to approximately 42 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
Number analyzed (Participants) | 143 | 146
Percentage of Participants | 90.9 [84.96 to 95.07] | 91.1 [85.26 to 95.17]

ADVERSE EVENTS:
Time Frame: Up to approximately 48 months
Description: All-Cause Mortality (ACM): all randomized participants, Up to approximately 48 months. AEs: All AEs were treatment-emergent AEs (TEAEs), defined as any AE which either began or worsened in severity on or after the date/time of first dose of study treatment and on or before 60 days after the date/time of last dose of study treatment.
Arm/Group | Placebo Combine With Chemotherapy | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy
All-Cause Mortality (participants affected / at risk) | 67/143 | 47/146
Serious Adverse Events (participants affected / at risk) | 62/143 | 64/146
Other Adverse Events (participants affected / at risk) | 143/143 | 146/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Combine With Chemotherapy (N=143) | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy (N=146)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 39 | 39
Infections and infestations (Infections and infestations) | 10 | 19
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 | 7
General disorders and administration site (General disorders) | 5 | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 2 | 6
Hepatobiliary disorders (Hepatobiliary disorders) | 4 | 5
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 2 | 4
Investigations (Investigations) | 3 | 1
Nervous system disorders (Nervous system disorders) | 3 | 4
Cardiac disorders (Cardiac disorders) | 1 | 2
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 3
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 1
Renal and urinary disorders (Renal and urinary disorders) | 1 | 3
Endocrine disorders (Endocrine disorders) | 0 | 2
psychiatric disorders (Psychiatric disorders) | 2 | 0
eye disorders (Eye disorders) | 0 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Combine With Chemotherapy (N=143) | TORIPALIMAB INJECTION(JS001 )Combine With Chemotherapy (N=146)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 142 | 143
Gastrointestinal disorders (Gastrointestinal disorders) | 138 | 135
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 118 | 116
Investigations (Investigations) | 91 | 88
General disorders and administration site conditions (General disorders) | 91 | 89
Nervous system disorders (Nervous system disorders) | 78 | 84
Respiratory, thoracic and mediastinal disorders Cough (Respiratory, thoracic and mediastinal disorders) | 71 | 69
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 50 | 68
Infections and infestations (Infections and infestations) | 38 | 62
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 40 | 43
Endocrine disorders (Endocrine disorders) | 27 | 53
Psychiatric disorders (Psychiatric disorders) | 30 | 37
Ear and labyrinth disorders (Ear and labyrinth disorders) | 18 | 22
Renal and urinary disorders (Renal and urinary disorders) | 10 | 18
Hepatobiliary disorders (Hepatobiliary disorders) | 7 | 12
Eye disorders (Eye disorders) | 7 | 12
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 | 8
Vascular disorders (Vascular disorders) | 21 | 32
Cardiac disorders (Cardiac disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03581786/Prot_SAP_ICF_000.pdf